CLINICAL TRIAL: NCT02394834
Title: An Exploratory Study of Treatment Sensitivity and Prognostic Factors in a Phase III, Randomized, Controlled Study Comparing the Efficacy and Safety of mFOLFOX6 + Bevacizumab Therapy vs. mFOLFOX6 + Panitumumab Therapy in Patients With Chemotherapy-naïve Wild-type RAS(KRAS/NRAS) Unresectable Advanced or Recurrent Colorectal Cancer
Brief Title: An Exploratory Study of Treatment Sensitivity and Prognostic Factors in a Efficacy and Safety Study of mFOLFOX6 + Bevacizumab Versus mFOLFOX6 + Panitumumab Therapy in Patients With Chemotherapy-naïve Unresectable Advanced or Recurrent Colorectal Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Panitumumab-4004; U1111-1167-3521 (Other: WHO); jRCT1080222785 (Registry Identifier: jRCT); UMIN000016782 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Metastatic colorectal cancer, Panitumumab, mFOLFOX6, Bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Panitumumab; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P; mFOLFOX6 + panitumumab combination therapy: OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 panitumumab: 6 mg/kg mFOLFOX6 + panitumumab combination therapy, once every two weeks
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab
- Group B; mFOLFOX6 + bevacizumab combination therapy: OXA: 85 mg/m2/day 1 l-LV: 200 mg/m2/day 1 5-FU iv: 400 mg/m2/day 1 5-FU civ: 2400 mg/m2/day 1-3 bevacizumab: 5 mg/kg/ mFOLFOX6 + bevacizumab combination therapy, once every two weeks
  Interventions: Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, bevacizumab

INTERVENTIONS:
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, panitumumab — oxaliplatin (OXA), levofolinate calcium (l-LV), panitumumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Groups: Group P; mFOLFOX6 + panitumumab combination therapy
Drug: oxaliplatin (OXA), levofolinate calcium (l-LV), 5-FU, bevacizumab — oxaliplatin (OXA), levofolinate calcium (l-LV), bevacizumab: intra-venous infusion 5-FU: bolus and continuous intra-venous infusion
  Groups: Group B; mFOLFOX6 + bevacizumab combination therapy

SUMMARY:
The purpose of this study is to investigate biomarkers which may be predictors of efficacy and safety of treatment with mFOLFOX6 + bevacizumab versus mFOLFOX6 + panitumumab therapy in patients with chemotherapy-naïve unresectable advanced or recurrent colorectal cancer.

DETAILED DESCRIPTION:
The drug being tested in this study is called Panitumumab. This exploratory study will investigate biomarkers which may be predictors of efficacy and safety of treatment with mFOLFOX6 + bevacizumab versus mFOLFOX6 + panitumumab therapy in patients with chemotherapy-naïve unresectable advanced or recurrent colorectal cancer.

Tumor tissue samples obtained from the participants who enrolled in the safety/efficacy study of Panitumumab + mFOLFOX versus bevacizumab + mFOLFOX (PARADIGM Study: NCT02394795) and provided consent for this additional study will be used. Mutations, amplification and rearrangement of predefined tumor-associated genes will be investigated using DNA collected from tumor samples used for assessing RAS mutations and plasma free DNA collected before administration of cycle 1 and at the discontinuation of the protocol treatment in the main study.

ELIGIBILITY:
Inclusion Criteria:

(1) Patients who are enrolled in the main study and personally provided written consent after adequately explained about the contents of the additional study

Exclusion Criteria:

(1) Patients who are determined by the investigator or researchers to be not suitable for participating in the additional study

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are enrolled in the main study and personally provided written consent after adequately explained about the contents of the additional study.
Sampling Method: Non-Probability Sample
Enrollment: 757 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 63 months
  OS obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between OS and gene mutations. OS will be measured as the time from the date of randomization to the date of death due to any causes.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 63 months
  PFS obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations. PFS is defined as the time from the date of randomization to the earlier of Progressive Disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or death due to any cause.
Response Rate (RR) | Approximately 12 months
  RR obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations. RR is defined as percentage of participants who achieve Complete Response (CR) and Partial Response (PR) as the best overall response per RECIST version 1.1.
Duration of Response (DOR) | Up to approximately 63 months
  DOR obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations. DOR means that the period from the day when either CR or PR is first confirmed until the day of documented PD or the day of death due to all causes, whichever occurs earlier.
Percentage of Participants who Proceeded to Surgical Resection | Up to approximately 63 month
  The outcome obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations.
Percentage of Participants with Early Tumor Shrinkage | Up to approximately 63 months
  The outcome obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations.
Degree of the Maximum Tumor Shrinkage (Depth of Response) | Up to approximately 63 months
  The outcome obtained in the main study will be stratified by the presence or absence of mutation of tumor-associated genes in tumor tissues at the baseline of the main study to evaluate the relationship between the efficacy endpoint and gene mutations.
Evaluation of the Relationship of Each Biomarker in Plasma Free DNA and Tumor Samples at Baseline of the Main Study | Up to approximately 63 months
Evaluation of the Relationship between Each Biomarker in Plasma Free DNA at Baseline of the Main Study, and Efficacy Endpoints | Up to approximately 63 months
Evaluation of the Relationship between a Change in Each Biomarker in Plasma Free DNA at Baseline and the Discontinuation of the Protocol Treatment of the Main Study, and Efficacy Endpoints | Up to approximately 63 months
Evaluation of the Relationship between a Change in Each Biomarker in Tumor Tissue at Baseline and the Discontinuation of the Protocol Treatment of the Main Study, and Efficacy Endpoints | Up to approximately 63 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (150):
- Japan (150):
  - Ichinomiya, Aichi-ken
  - Komaki, Aichi-ken
  - Kounan, Aichi-ken
  - Nagakute, Aichi-ken
  - Nagoya, Aichi-ken
  - Okazaki, Aichi-ken
  - Toyohashi, Aichi-ken
  - Toyokawa, Aichi-ken
  - Toyota, Aichi-ken
  - Yatomi, Aichi-ken
  - Daisen, Akita
  - Hirosaki, Aomori
  - Misawa, Aomori
  - Kashiwa, Chiba
  - Yachiyo, Chiba
  - Matsuyama, Ehime
  - Tōon, Ehime
  - Tsuruga, Fukui
  - Yoshida, Fukui
  - Kitakyushu, Fukuoka
  - Koga, Fukuoka
  - Kurume, Fukuoka
  - Omuta, Fukuoka
  - Aizu-Wakamatsu, Fukushima
  - Iwaki, Fukushima
  - Kōriyama, Fukushima
  - Shirakawa, Fukushima
  - Hashima, Gifu
  - Kakamigahara, Gifu
  - Minokamo, Gifu
  - Okazai, Gifu
  - Ōgaki, Gifu
  - Maebashi, Gunma
  - Ōta, Gunma
  - Fukuyama, Hiroshima
  - Hakodate, Hokkaido
  - Kitami, Hokkaido
  - Kushiro, Hokkaido
  - Obihiro, Hokkaido
  - Otaru, Hokkaido
  - Sapporo, Hokkaido
  - Akashi, Hyōgo
  - Amagasaki, Hyōgo
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Nishinomiya, Hyōgo
  - Hitachi, Ibaraki
  - Kasama, Ibaraki
  - Ryūgasaki, Ibaraki
  - Tsuchiura, Ibaraki
  - Tsukuba, Ibaraki
  - Hakusan, Ishikawa-ken
  - Kaga, Ishikawa-ken
  - Kahoku, Ishikawa-ken
  - Kanazawa, Ishikawa-ken
  - Nanao, Ishikawa-ken
  - Morioka, Iwate
  - Kida, Kagawa-ken
  - Marugame, Kagawa-ken
  - Takamatsu, Kagawa-ken
  - Fujisawa, Kanagawa
  - Hiratsuka, Kanagawa
  - Isehara, Kanagawa
  - Kamakura, Kanagawa
  - Kanazawachō, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Yokosuka, Kanagawa
  - Nankoku, Kochi
  - Matsuzaka, Mie-ken
  - Tsu, Mie-ken
  - Yokkaichi, Mie-ken
  - Ishinomaki, Miyagi
  - Murata, Miyagi
  - Natori-shi, Miyagi
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Saku, Nagano
  - Ōmura, Nagasaki
  - Sasebo, Nagasaki
  - Ikoma, Nara
  - Tenri, Nara
  - Yamatotakada, Nara
  - Yufu, Oita Prefecture
  - Kurashiki, Okayama-ken
  - Naha, Okinawa
  - Tomigusuku, Okinawa
  - Urasoe, Okinawa
  - Hirakata, Osaka
  - Kawachi-Nagano, Osaka
  - Moriguchi, Osaka
  - Neyagawa, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Kawagoe, Saitama
  - Kitaadachi, Saitama
  - Koshigaya, Saitama
  - Moriyama, Shiga
  - Ōtsu, Shiga
  - Izumi, Shimane
  - Izumo, Shimane
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Sunto, Shizuoka
  - Shimotsuga, Tochigi
  - Shimotsuke, Tochigi
  - Utsunomiya, Tochigi
  - Komatsushimachō, Tokushima
  - Bunkyo-ku, Tokyo
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Koto-ku, Tokyo
  - Machida, Tokyo
  - Minato-ku, Tokyo
  - Musashino, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjyuku-ku, Tokyo
  - Yonago, Tottori
  - Kurobe-shi, Toyama
  - Takaoka, Toyama
  - Sakata, Yamagata
  - Tsuruoka, Yamagata
  - Iwakuni, Yamaguchi
  - Kofu, Yamanashi
  - Akita
  - Aomori
  - Chiba
  - Fukui
  - Fukuoka
  - Gifu
  - Kagoshima
  - Kochi
  - Kumamoto
  - Kyoto
  - Miyazaki
  - Nagano
  - Nagasaki
  - Niigata
  - Okayama
  - Okinawa
  - Osaka
  - Saga
  - Saitama
  - Shizuoka
  - Tokushima
  - Toyama
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Shitara K, Muro K, Watanabe J, Yamazaki K, Ohori H, Shiozawa M, Takashima A, Yokota M, Makiyama A, Akazawa N, Ojima H, Yuasa Y, Miwa K, Yasui H, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Mori I, Yamanaka K, Hihara M, Soeda J, Misumi T, Yamamoto K, Yamashita R, Akagi K, Ochiai A, Uetake H, Tsuchihara K, Yoshino T. Baseline ctDNA gene alterations as a biomarker of survival after panitumumab and chemotherapy in metastatic colorectal cancer. Nat Med. 2024 Mar;30(3):730-739. doi: 10.1038/s41591-023-02791-w. Epub 2024 Feb 12. PMID 38347302
- [Derived] Yoshino T, Uetake H, Tsuchihara K, Shitara K, Yamazaki K, Oki E, Sato T, Naitoh T, Komatsu Y, Kato T, Yamanaka K, Iwasaki K, Soeda J, Hihara M, Yamanaka T, Ochiai A, Muro K. Rationale for and Design of the PARADIGM Study: Randomized Phase III Study of mFOLFOX6 Plus Bevacizumab or Panitumumab in Chemotherapy-naive Patients With RAS (KRAS/NRAS) Wild-type, Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2017 Jun;16(2):158-163. doi: 10.1016/j.clcc.2017.01.001. Epub 2017 Jan 24. PMID 28237539
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b60294db2bf003ab499d5